CLINICAL TRIAL: NCT05466370
Title: Prediction of Transfusion-Associated Complications
Acronym: PRETRACO
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PRETRACO
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Transfusion-dependent Anemia
Keywords: Artificial Intelligence; Machine Learning; Transfusion; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AKI: Acute Kidney Injury
  Interventions: Biological: Transfusion of Allogeneic Blood
- ARF: Acute Respiratory Failure
  Interventions: Biological: Transfusion of Allogeneic Blood
- AKI and ARF: Acute Kidney Injury and Acute Respiratory Failure
  Interventions: Biological: Transfusion of Allogeneic Blood
- no complication: no complication
  Interventions: Biological: Transfusion of Allogeneic Blood

INTERVENTIONS:
Biological: Transfusion of Allogeneic Blood — Transfusion of Allogeneic Blood

SUMMARY:
Currently, about 350000 red blood cell concentrates are produced from blood donations in Austria every year.

In addition to the main effect of replacing lost blood, red blood cell concentrates also have many undesirable effects - from blood group compatibilities, which are easily avoidable due to care, to storage-related side effects, to mostly intensive care problems as a result of massive transfusions, to system-wide effects such as TRALI, TACO and TRIM.

Before being administered to patients, red blood cell concentrates undergo an extensive quality assurance process in which a large number of parameters are collected. Prior to use on patients, for example, bedside tests and tests for further incompatibilities with a blood sample from the intended patient are performed. With the implementation of Patient Blood Management (PBM) in recent years, the use of red cell concentrates has become more targeted - the number of transfusions is decreasing in most developed countries. However, it is still possible to suffer transfusion-related adverse events (TRAE). Thus, active research activity to reduce these TRAEs continues to be called for.

To date, however, it is not known which patients experience transfusion-related adverse events. Despite the broad measures of hemovigilance and pre-transfusion testing, it is still not possible to predict which individual patient will respond to a transfusion with a typical adverse event such as hypotension, hemolysis, renal failure, or TRALI. It seems understandable that characteristics of the patient as well as characteristics of the administered unit could play a role for this. In particular, it is conceivable that a combination of characteristics of the blood unit and characteristics of the patient could determine a complication in the course of administration. For this reason, it seems attractive to use artificial intelligence and machine learning methods to predict any complications.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients that received at a blood transfusion the Kepler University Hospital in the period between 2016-10-31 to 2020-08-31.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As described in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3366 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
AUROC for Classification of AKI | 2016-10-31 to 2020-08-31
  AUROC for Classification of AKI
AUROC for Classification of ARF | 2016-10-31 to 2020-08-31
  AUROC for Classification of ARF
AUROC for Classification of AKI and ARF | 2016-10-31 to 2020-08-31
  AUROC for Classification of AKI and ARF

SECONDARY OUTCOMES:
Confusion Matrix | 2016-10-31 to 2020-08-31
  Confusion Matrix Results: true positives, true negatives, false positive, false negatives and values calculated from these results.
Descriptive Statistics | 2016-10-31 to 2020-08-31
  Descriptive Statistics (age in years, gender as male/female, blood group as A, B, 0, AB, hemoglobin in g/dl, platelets in count/microliter, leukocytes in cells per liter, CRP in mg/dl, creatinine in mg/dl, GFR ml/minute, glucose in mg/dl, potassium in mmol/l, TT, aPTT in seconds, ALT U/liter, paO2 mmHg, Rhesus type as positive or negative, height in cm, weight in kg, body temperature in kg, age of blood in days, cholesterine in mg/dl, systolic blood pressure in mmHg, diastolic blood pressure in mmHg)
  This outcome measure will compare the individual feature (e. g. height in cm) in one group vs. the other. Significant difference will be described by p-value.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tschoellitsch, MD, Principal Investigator — Kepler University Hospital and Johannes Kepler University, Linz, Austria
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschoellitsch T, Moser P, Maletzky A, Seidl P, Bock C, Roland T, Ludwig H, Sussner S, Hochreiter S, Meier J. Potential Predictors for Deterioration of Renal Function After Transfusion. Anesth Analg. 2024 Mar 1;138(3):645-654. doi: 10.1213/ANE.0000000000006720. Epub 2024 Feb 16. PMID 38364244